CLINICAL TRIAL: NCT01202864
Title: Ethnic/Racial Variations of Intracerebral Hemorrhage (ERICH)
Acronym: ERICH
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Massachusetts General Hospital (Other); Columbia University (Other); University of Maryland (Other); Georgetown University (Other); Wake Forest University (Other); Emory University (Other); University of Miami (Other); University of Illinois at Chicago (Other); University of Texas, Southwestern Medical Center at Dallas (Other); The University of Texas Health Science Center, Houston (Other); The University of Texas Health Science Center at San Antonio (Other); University of New Mexico (Other); University of Arizona (Other); University of Southern California (Other); St. Luke's-Roosevelt Hospital Center (Other); University of California, San Francisco (Other); Duke University (Other); University of Virginia (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Daniel Woo, Professor, University of Cincinnati
Other Study IDs: 1008059; R01NS069763-01 (Other Grant/Funding Number: NINDS)
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; ICH; Stroke; Cerebrovascular accident
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: 3000 Cases
- Controls: 3000 Controls

SUMMARY:
The purpose of this study is to find risk factors for hemorrhagic stroke, specifically intracerebral hemorrhage (ICH), among Caucasians, African Americans, and Hispanics.

ELIGIBILITY:
Inclusion Criteria:

All cases must meet the following eligibility criteria:

1. Age 18 years or greater, fulfillment of the criteria for intracerebral hemorrhage
2. Resident for at least 6 months within 50 miles of the recruiting center
3. No evidence of trauma, vascular malformation or aneurysm, or brain tumor as a cause of the hemorrhage
4. Ability of the patient or legal representative to provide informed consent

Exclusion Criteria:

Exclusion Criteria:

1. Malignancies leading to coagulopathy
2. Hemorrhagic transformation of ischemic infarct
3. Hemorrhage secondary to dural venous sinus thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our purpose is to enroll 1000 cases of ICH among whites, 1000 cases of ICH among blacks, and 1000 cases of ICH among Hispanics.
  3000 controls matched to cases by race/ethnicity, age (+/- 5 years), gender, and geographic location.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Woo, MD, MS, Principal Investigator — University of Cincinnati; Matthew Flaherty, MD, Principal Investigator — University of Cincinnati
Locations (15):
- United States (15):
  - University of Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Miami - Biorepository, Miami, Florida
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Medical School at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Taylor TN, Davis PH, Torner JC, Holmes J, Meyer JW, Jacobson MF. Lifetime cost of stroke in the United States. Stroke. 1996 Sep;27(9):1459-66. doi: 10.1161/01.str.27.9.1459. PMID 8784113
- [Background] Woo D, Sauerbeck LR, Kissela BM, Khoury JC, Szaflarski JP, Gebel J, Shukla R, Pancioli AM, Jauch EC, Menon AG, Deka R, Carrozzella JA, Moomaw CJ, Fontaine RN, Broderick JP. Genetic and environmental risk factors for intracerebral hemorrhage: preliminary results of a population-based study. Stroke. 2002 May;33(5):1190-5. doi: 10.1161/01.str.0000014774.88027.22. PMID 11988589
- [Background] Kissela B, Schneider A, Kleindorfer D, Khoury J, Miller R, Alwell K, Woo D, Szaflarski J, Gebel J, Moomaw C, Pancioli A, Jauch E, Shukla R, Broderick J. Stroke in a biracial population: the excess burden of stroke among blacks. Stroke. 2004 Feb;35(2):426-31. doi: 10.1161/01.STR.0000110982.74967.39. PMID 14757893
- [Background] Hardie K, Hankey GJ, Jamrozik K, Broadhurst RJ, Anderson C. Ten-year survival after first-ever stroke in the perth community stroke study. Stroke. 2003 Aug;34(8):1842-6. doi: 10.1161/01.STR.0000082382.42061.EE. Epub 2003 Jul 3. PMID 12843343
- [Background] Broderick JP, Phillips SJ, Whisnant JP, O'Fallon WM, Bergstralh EJ. Incidence rates of stroke in the eighties: the end of the decline in stroke? Stroke. 1989 May;20(5):577-82. doi: 10.1161/01.str.20.5.577. PMID 2718196
- [Background] Broderick JP, Brott T, Tomsick T, Miller R, Huster G. Intracerebral hemorrhage more than twice as common as subarachnoid hemorrhage. J Neurosurg. 1993 Feb;78(2):188-91. doi: 10.3171/jns.1993.78.2.0188. PMID 8421201
- [Background] Barber M, Stott DJ. Validity of the Telephone Interview for Cognitive Status (TICS) in post-stroke subjects. Int J Geriatr Psychiatry. 2004 Jan;19(1):75-9. doi: 10.1002/gps.1041. PMID 14716702
- [Background] de Jager CA, Budge MM, Clarke R. Utility of TICS-M for the assessment of cognitive function in older adults. Int J Geriatr Psychiatry. 2003 Apr;18(4):318-24. doi: 10.1002/gps.830. PMID 12673608
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] RANKIN J. Cerebral vascular accidents in patients over the age of 60. II. Prognosis. Scott Med J. 1957 May;2(5):200-15. doi: 10.1177/003693305700200504. No abstract available. PMID 13432835
- [Background] Flibotte JJ, Hagan N, O'Donnell J, Greenberg SM, Rosand J. Warfarin, hematoma expansion, and outcome of intracerebral hemorrhage. Neurology. 2004 Sep 28;63(6):1059-64. doi: 10.1212/01.wnl.0000138428.40673.83. PMID 15452298
- [Background] Goldstein JN, Fazen LE, Snider R, Schwab K, Greenberg SM, Smith EE, Lev MH, Rosand J. Contrast extravasation on CT angiography predicts hematoma expansion in intracerebral hemorrhage. Neurology. 2007 Mar 20;68(12):889-94. doi: 10.1212/01.wnl.0000257087.22852.21. PMID 17372123
- [Background] Kumar MA, Rost NS, Snider RW, Chanderraj R, Greenberg SM, Smith EE, Rosand J. Anemia and hematoma volume in acute intracerebral hemorrhage. Crit Care Med. 2009 Apr;37(4):1442-7. doi: 10.1097/CCM.0b013e31819ced3a. PMID 19242340
- [Background] Brott T, Broderick J, Kothari R, Barsan W, Tomsick T, Sauerbeck L, Spilker J, Duldner J, Khoury J. Early hemorrhage growth in patients with intracerebral hemorrhage. Stroke. 1997 Jan;28(1):1-5. doi: 10.1161/01.str.28.1.1. PMID 8996478
- [Background] Davis SM, Broderick J, Hennerici M, Brun NC, Diringer MN, Mayer SA, Begtrup K, Steiner T; Recombinant Activated Factor VII Intracerebral Hemorrhage Trial Investigators. Hematoma growth is a determinant of mortality and poor outcome after intracerebral hemorrhage. Neurology. 2006 Apr 25;66(8):1175-81. doi: 10.1212/01.wnl.0000208408.98482.99. PMID 16636233
- [Background] Mayer SA, Brun NC, Begtrup K, Broderick J, Davis S, Diringer MN, Skolnick BE, Steiner T; FAST Trial Investigators. Efficacy and safety of recombinant activated factor VII for acute intracerebral hemorrhage. N Engl J Med. 2008 May 15;358(20):2127-37. doi: 10.1056/NEJMoa0707534. PMID 18480205
- [Derived] Behymer TP, Sekar P, Demel SL, Aziz YN, Coleman ER, Williamson BJ, Stanton RJ, Sawyer RP, Turner AC, Vagal VS, Osborne J, Gilkerson LA, Comeau ME, Flaherty ML, Langefeld CD, Woo D. Psychosocial Stress and Risk for Intracerebral Hemorrhage in the ERICH (Ethnic/Racial Variations of Intracerebral Hemorrhage) Study. J Am Heart Assoc. 2025 Mar 18;14(6):e024457. doi: 10.1161/JAHA.121.024457. Epub 2025 Mar 7. PMID 40055853
- [Derived] Ridha M, Hannawi Y, Murthy S, Carvalho Poyraz F, Kumar A, Park S, Roh D, Sekar P, Woo D, Burke J. Premorbid Blood Pressure Control Modifies Risk of DWI Lesions With Acute Blood Pressure Reduction in Intracerebral Hemorrhage. Hypertension. 2024 Oct;81(10):2113-2123. doi: 10.1161/HYPERTENSIONAHA.124.23271. Epub 2024 Jul 29. PMID 39069917
- [Derived] Ng Y, Qi W, King NKK, Christianson T, Krishnamoorthy V, Shah S, Divani A, Bettin M, Coleman ER, Flaherty ML, Walsh KB, Testai FD, McCauley JL, Gilkerson LA, Langefeld CD, Behymer TP, Woo D, James ML. Initial antihypertensive agent effects on acute blood pressure after intracerebral haemorrhage. Stroke Vasc Neurol. 2022 Oct;7(5):367-374. doi: 10.1136/svn-2021-001101. Epub 2022 Apr 20. PMID 35443984
- [Derived] Liu L, Fuller M, Behymer TP, Ng Y, Christianson T, Shah S, King NKK, Woo D, James ML. Selective Serotonin Reuptake Inhibitors and Intracerebral Hemorrhage Risk and Outcome. Stroke. 2020 Apr;51(4):1135-1141. doi: 10.1161/STROKEAHA.119.028406. Epub 2020 Mar 4. PMID 32126942
- [Derived] James ML, Langefeld CD, Sekar P, Moomaw CJ, Elkind MSV, Worrall BB, Sheth KN, Martini SR, Osborne J, Woo D; ERICH Investigators. Assessment of the interaction of age and sex on 90-day outcome after intracerebral hemorrhage. Neurology. 2017 Sep 5;89(10):1011-1019. doi: 10.1212/WNL.0000000000004255. Epub 2017 Jul 14. PMID 28710330
- [Derived] Walsh KB, Woo D, Sekar P, Osborne J, Moomaw CJ, Langefeld CD, Adeoye O. Untreated Hypertension: A Powerful Risk Factor for Lobar and Nonlobar Intracerebral Hemorrhage in Whites, Blacks, and Hispanics. Circulation. 2016 Nov 8;134(19):1444-1452. doi: 10.1161/CIRCULATIONAHA.116.024073. Epub 2016 Oct 13. PMID 27737957